CLINICAL TRIAL: NCT06139016
Title: Using Virtual Reality to Control the Audio-visual Inputs During Ketamine/Esketamine Treatment
Acronym: VR-KET
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000036184; 000 (Other: CTGTY)
Record Dates: First submitted 2023-11-03; First posted 2023-11-18 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Depression
Keywords: ketamine; esketamine; virtual reality
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment group (Experimental): This single arm will include all participants of the study, who will all receive the intervention
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — Virtual reality gear and content will be used to affect and control the audiovisual perception of patients during a single treatment with ketamine/esketamine

SUMMARY:
Investigators aim to examine the role of audiovisual inputs during treatment with ketamine/esketamine in affecting tolerability and effectiveness of treatment of depressive episodes, by providing patients with a relaxing environment using virtual reality goggles and noise cancelling headphones, and assessing whether these tools can improve the tolerability and effectiveness of treatment with ketamine/esketamine

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years old
* Patients must have completed the acute series of treatment and weekly optimization phases of ketamine/esketamine treatment, and currently receiving continuation/maintenance treatment Written consent for the study procedures
* Ability and willingness, in the investigator's judgement, to comply with the study procedure and study requirements.

Exclusion Criteria:

* Hearing or visual impairment to the degree that would interfere with ability to see or hear VR content.
* Difficulty in understanding spoken or written English
* Unable to provide informed consent
* Dementia or other cognitive disorder or intellectual disability that would impair the subject's ability to understand the study procedure (per investigator judgment)
* Any other medical or psychiatric comorbidity that the investigator judges would put the participant at additional undue risk due to study participation or would impair subject's ability to participate in the study.
* Was previously enrolled/randomized into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Tolerability of VR treatment assessed by qualitative report | baseline and Immediately post-VR treatment
  Tolerability of VR treatment will be assessed by qualitative report, an open-ended question where the participant is allowed to describe any concerns not covered by SAFTEE assessment.
Safety of VR treatment assessed by Systematic Assessment of Treatment Emergent Events (SAFTEE) assessment | baseline, during VR treatment and Immediately post-VR treatment
  The SAFTEE assessment will be used to assess adverse events during the trial by the number of participants that had any adverse events while on study.
Change in overall treatment experience satisfaction between the pre-VR and VR treatment sessions | Baseline and immediately post VR treatment session
  Efficacy will be assessed by the difference in overall treatment experience satisfaction (via Likert scale) between the pre-VR and VR treatment sessions. Total scores range from 0 to 10 with higher scores indicating higher satisfaction with the treatment experience.

SECONDARY OUTCOMES:
Change in 5-Dimensional Altered States of Consciousness Questionnaire (5D-ASC) subscale scores | baseline, during VR treatment and Immediately post-VR treatment
  The 5D-ASC measures altered states of consciousness and contains 94 items using visual analogue scales. Score for each will be calculated from 0 to 100 based on measurement of where the participant has drawn the line. Then each subscale is the median score from a pre-defined list of items (eg subscale 2 is median of items 9,81,94). Higher scores means more altered state of consciousness.
Change in 5D-ASC total score | baseline, during VR treatment and Immediately post-VR treatment
  The 5D-ASC measures altered states of consciousness and contains 94 items (visual analogue scales. Score for each will be calculated from 0 to 100 based on measurement of where the participant has drawn the line. Total score is the median of all items. Higher scores means more altered state of consciousness.
Change in The Clinician-Administered Dissociative States Scale (CADSS) | baseline, 40 minutes and immediately post VR treatment
  The CADSS is a 23 item structured clinical interview to assess state dissociation rated by clinicians. Each item is scored from 0 (not at all) to 4 (extreme). Total score range from 0-92 with higher scores indicating greater severity of dissociative experiences.
Change in participant experience | baseline, during VR treatment and Immediately post-VR treatment
  Participant experience will be assessed by self report on whether it was a "pleasant vs unpleasant experience"using a Likert scale. Scores from 0-11 with higher scores indicating a more pleasant experience.
Change in level of relaxation | baseline, during VR treatment and Immediately post-VR treatment
  The "level of relaxation" will be scored using a Likert scale with total score range from 0 to 11. Higher scores indicate a higher level of relaxation.

CONTACTS AND LOCATIONS:
Overall Officials: Sina Nikayin, MD, Principal Investigator — Assistant Professor, Departement of Psychiatry, Yale University
Locations (1):
- Yale Psychiatry Hospital Interventional Psychiatry Services (IPS) unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No